CLINICAL TRIAL: NCT01798043
Title: Impact of Septal Vs Apical Pacing on Right and Left Ventricular Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow enrolment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-12-048-CH-LV
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Heart Block; Sick Sinus Syndrome; Atrioventricular Block; Ventricular Dysfunction
MeSH Terms: conditions — Heart Block; Sick Sinus Syndrome; Atrioventricular Block; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Septal RV lead with >50% pacing (B1) (Experimental): Cardiac MRI with pacemaker stimulation
  Interventions: Other: Cardiac MRI with pacemaker stimulation
- Septal RV lead with <50% pacing (B2) (Experimental): Cardiac MRI with and without pacemaker stimulation
  Interventions: Other: Cardiac MRI with and without pacemaker stimulation
- Apical RV lead with >50% pacing (A1) (Experimental): Cardiac MRI with pacemaker stimulation
  Interventions: Other: Cardiac MRI with pacemaker stimulation
- Apical RV lead with <50% pacing (A2) (Experimental): Cardiac MRI with and without pacemaker stimulation
  Interventions: Other: Cardiac MRI with and without pacemaker stimulation

INTERVENTIONS:
Other: Cardiac MRI with pacemaker stimulation — Patient is undergoing a Cardiac MRI at enrollment and 12 months later
  Arms: Apical RV lead with >50% pacing (A1); Septal RV lead with >50% pacing (B1)
Other: Cardiac MRI with and without pacemaker stimulation — Patient is undergoing a Cardiac MRI at enrollment and 12 months later
  Arms: Apical RV lead with <50% pacing (A2); Septal RV lead with <50% pacing (B2)

SUMMARY:
The study aims to use cardiac MRI scans and analysis techniques to evaluate differences in cardiac function after 12 months of pacing in patients with pacing leads placed in different positions within the right ventricle (apically or septally).

DETAILED DESCRIPTION:
Prolonged pacing from the right ventricular (RV) Apex has been shown to be associated with progressive left ventricular (LV) dysfunction. This has led to an interest in alternative right ventricular pacing sites. Only very few studies investigated the effect of alternative right ventricular pacing sites using three dimensional imaging. Using cardiac MRI volumetric left- and right ventricular analysis and three-dimensional reconstruction is more accurate compared to trans-thoracic echocardiogram. St. Jude Medical has developed a MRI conditional pacemaker system enabling for the first time to investigate alternative pacing sites using cardiac MRI.

Patients already implanted with an MRI conditional pacemaker system from St. Jude Medical will be enrolled in that study and subdivided into 4 groups (right ventricular pacing lead positioned apically or septally subdivided in patients paced for <50% of time or 50% or more). All patients will undergo cardiac MRI at enrollment and again 12 months later. Patients paced <50% of the time will undergo cardiac MRI with and without pacemaker stimulation at both visits.

ELIGIBILITY:
Inclusion Criteria:

* Have been implanted with an Accent MRI pacemaker and Tendril MRI leads.
* Have an RV lead implanted apically (group A) or septally (Group B)
* Are RV paced for <50% of the time (groups A2 and B2)
* Are RV paced for > 50% of the time (Groups A1 and B1)
* Are ≥ 18 years of age.
* Are able to provide written informed consent.
* Are willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

* Have permanent atrial fibrillation with preserved intrinsic conduction
* Have a non-MRI compatible device or material implant (e.g., intracranial aneurysm clip, non-MRI compatible devices or material, metals or alloys, etc.).
* Have a lead extender, plug or adaptor.
* Do not have an RV lead implanted apically or septally.
* Are eligible for groups A1 or B1 but appropriate group already has 20 patients enrolled.
* Are eligible for groups A2 or B2 but appropriate group already has 5 patients enrolled
* Are currently participating in another device or drug investigation which includes an active treatment arm.
* Are pregnant or planning to become pregnant during the duration of the study.
* Have a life expectancy of less than 12 months from Screening due to any life-threatening condition.
* Are contraindicated for an MRI scan due to any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in LV chamber volumes. | 12 months (baseline to end of study)

SECONDARY OUTCOMES:
Change in Dyssynchrony | 12 months
Change in Ejection fraction | 12 months
Change in Strain rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Zbinden, MD, Principal Investigator — Triemli Hospital
Locations (1):
- Stadtspital Triemli, Zurich, Switzerland